CLINICAL TRIAL: NCT07265609
Title: A Two-year Comparative Evaluation of Clinical Performance of a CAD/CAM Composite to a Polymer-infiltrated Ceramic Restorations
Brief Title: Clinical Performance of Two Different Resin-Matrix Ceramic Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: J0022055023CD
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dental Restoration Failure
Keywords: Resin-matrix ceramics; Polymer-infiltrated ceramics; Resin nano-ceramics; Indirect restorations; CAD/CAM
MeSH Terms: interventions — Inlays

STUDY DESIGN:
Intervention Model Description: The study is a randomized split-mouth clinical trial. Each participant received both restorative materials: a resin-nanoceramic and a polymer-infiltrated ceramic. Randomization assigned one material to one side of the mouth and the other material to the contralateral side for each participant. Treatments were applied according to the manufacturers' instructions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin nano-ceramic (Active Comparator): Resin-matrix ceramic CAD/CAM blocks for indirect restorations. Restorations were designed, milled, finished, and cemented on the assigned contralateral site according to the manufacturer's instructions. Each patient received this material on one side of the mouth; side allocation was randomized.
  Interventions: Other: inlays
- Polymer-infiltrated ceramics (Active Comparator): Resin-matrix ceramic CAD/CAM blocks for indirect restorations. Restorations were designed, milled, finished, and cemented on the assigned contralateral site according to the manufacturer's instructions. Each patient received this material on one side of the mouth; side allocation was randomized.
  Interventions: Other: inlays

INTERVENTIONS:
Other: inlays — Inlay cavity preparations were performed, and RMC restorations were designed, milled, finished, and cemented on the assigned contralateral site according to the manufacturer's instructions. Each patient received one material on one side of the mouth and the other on the contralateral side. Side allocation was randomized.
  Other Names: Indirect restorations; partial-coverage restorations

SUMMARY:
This study was designed to evaluate and compare the 2-year clinical performance of two different resin-matrix ceramic inlays

DETAILED DESCRIPTION:
The design of this prospective randomized controlled clinical trial was a split-mouth, two-arm, double-blinded clinical trial, with an allocation ratio of 1:1. The reporting of the trial followed the Consolidated Standards of Reporting Trials (CONSORT) Statement. Twelve adult patients seeking dental treatments in the Conservative Dentistry Department outpatient clinic, Faculty of Dentistry, Mansoura University, were enrolled in the current study with a total of twenty-four compound inlay cavities. Each patient must sign a consent form before participating in the current study. The study was conducted from August 2023 to August 2025 as a part of the doctoral dissertation. Mansoura University's institution's ethics committee approved the form and protocol before conducting the study. The sample size was calculated using the G*Power statistical program. Based on an effect size of 0.4, a significance level of 5% (p < 0.05), and a statistical power of 80%, a minimum of 10 samples per group was required. To compensate for potential dropouts, the total sample size was increased to 12 patients, yielding a total of 24 restorations.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of two molars with compound proximal carious lesions or defective restorations involving two surfaces (occluso-mesial or occluso-distal cavities) corresponding to Black's Class II, with a severity score of 4 or 5 according to the International Caries Detection and Assessment System (ICDAS)
2. The buccolingual width of lesions should exceed two-thirds of the intercuspal distance.
3. The teeth were required to be vital and free from any periapical radiolucency.
4. The teeth were required to be in normal alignment, in contact with sound adjacent teeth, and have antagonist teeth present in normal occlusion.

Exclusion Criteria:

1. The presence of uncontrolled systemic disease, pregnancy or breastfeeding.
2. Patients with extremely poor oral hygiene, active periodontal disease, or those involving in orthodontic treatment or periodontal surgery.
3. Patients with wear facets and parafunctional habits as clinching and bruxism.
4. Hypersensitive, endodontically treated, non-vital or cracked teeth.
5. Teeth with proximal cavities involving more than two surfaces, those that exhibited pulp exposure during caries excavation and required direct pulp capping, or those with missing cusps necessitating cusp capping.
6. Teeth without proximal contact, missing neighbouring or opposing teeth
7. Patients with known unavailability to attend recall visits, or with known allergy to any component of the study materials.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Esthetic, functional and biological properties for each CAD/CAM restorative material | 2 years
  Esthetic, functional and biological properties were assessed using World Dental Federation (FDI) criteria. Each criterion was rated on a five-point scale, where a score of 1 indicated clinically excellent or very good performance, score 2 indicated clinically good, score 3 indicated a clinically satisfactory, score 4 indicated clinically unsatisfactory, and score 5 indicated clinically poor performance requiring repair or replacement.

SECONDARY OUTCOMES:
Radiographic examination | 2 years
  Each material was examined radiographically and radiographs were assessed and rated following World Dental Federation (FDI) five-point scale, where a score of 1 indicated clinically excellent or very good performance, score 2 indicated clinically good, score 3 indicated a clinically satisfactory, score 4 indicated clinically unsatisfactory, and score 5 indicated clinically poor performance requiring repair or replacement.
Periodontal response and adjacent mucosa | 2 years
  Periodontal responce and adjacent mucosa were assessed using World Dental Federation (FDI) criteria. Each criterion was rated on a five-point scale, where a score of 1 indicated clinically excellent or very good performance, score 2 indicated clinically good, score 3 indicated a clinically satisfactory, score 4 indicated clinically unsatisfactory, and score 5 indicated clinically poor performance requiring repair or replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Fathy, Assistant Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt; Hamdi Hamama, Clinical Professor, Study Director — Faculty of Dentistry, Mansoura Universtity, Egypt; Jukka P Matinlinna, Clinical Professor, Study Director — School of Medical Science, University of Manchester, M13 9PL, Manchester, UK; Salah H Mahmoud, Clinical Professor, Study Chair — Faculty of Dentistry, Mansoura Universtity, Egypt
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months for 3 years
Access Criteria: for anyone